CLINICAL TRIAL: NCT03931369
Title: Single Administration of TOLVAptan at a Dosage Used in the Treatment of Hyponatremia: Changes in THIRST and Water Balance in Healthy Volunteers
Brief Title: Adaptation of Thirst to a Single Administration of Tolvaptan (TOLVATHIRST)
Acronym: TOLVATHIRST
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Otsuka Pharmaceutical Europe Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APHP180494; 2019-001335-31 (EudraCT Number)
Record Dates: First submitted 2019-04-15; First posted 2019-04-30 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tolvaptan test (Experimental): 15 MG pill administered tolvatan once, one day
  Interventions: Drug: Tolvaptan 15 MG

INTERVENTIONS:
Drug: Tolvaptan 15 MG — Single administration of one pill of 15 MG tolvaptan

SUMMARY:
Tolvaptan is a new drug that specifically antagonizes the V2-receptor of antidiuretic hormone (ADH) and leads to water diuresis: During acute administration of tolvaptan, the main fear is to induce a too fast increase in plasma sodium concentration and in turn brain damageHowever, the tolvaptan-induced increase in plasma sodium concentration is expected to stimulate thirst, preventing major negative water balance.

The investigators hypothesize that tolvaptan-induced increase in plasma osmolality (and sodium concentration) is dependent of thirst adaptation that is influenced by physiological factors, namely age and sex. To address the effect of a single oral administration of tolvaptan at a dosage used during hyponatremia (15 mg) under free water access in healthy volunteers. Primary outcome will be the maximal change in serum sodium concentration within the 6 hours following tolvaptan administration.

DETAILED DESCRIPTION:
Tolvaptan is a new drug that specifically antagonizes the V2-receptor of antidiuretic hormone (ADH) and leads to water diuresis: its beneficial effects have been demonstrated for hyponatremia due to a syndrome of inappropriate antidiuresis (SIAD). During acute administration of tolvaptan, the main fear is to induce a too fast increase in plasma sodium concentration and in turn brain damage. An acute increase in serum sodium concentration has been observed in water restricted subjects. However, the tolvaptan-induced increase in plasma sodium concentration is expected to stimulate thirst, preventing major negative water balance. In non-water restricted subjects, this has never been studied. Moreover, this physiological adaptation may change according to age and gender. The investigatorshypothesize that healthy volunteers will adapt normally to an acute tolvaptan administration, thirst helping to maintain plasma sodium and osmolality within the normal range. The final tolvaptan-induced increase in plasma osmolality will depend on thirst adaptation, influenced by physiological factors, namely age and sex.

Sixty subjects (30 male, 30 female) from 18 to 85 years old will be recruited from the database of healthy subjects of the Clinical Investigation Center of the European Georges Pompidou Hospital, Paris, France. They will have two visits: one inclusion safety visit without administration, and 2 to 15 days later, an experimental visit. During the later visit water and electrolyte output and water intake will be monitored hourly two hours before and six hours after single administration of 15 mg tolvaptan.

ELIGIBILITY:
Inclusion Criteria:

* To be 18-85 years old at the date of inclusion, both sex
* to have his/her full-legal capacity and understand the study protocol,
* to be covered by health insurance,
* to give his/her written informed consent

Exclusion Criteria:

* On-going pregnancy,
* women of childbearing age without efficient contraception,
* breastfeeding women,
* all acute (less than 7 days) pathological conditions,
* all active chronic diseases, especially those that could be interfering with water balance and/or thirst and/or renal response to tolvaptan,
* any prohibited treatment since at least 8 days (tolerated : calcium channel blockers, statins, acetaminophen, oral contraception and impregnated sterilets of progesterone are tolerated if necessary),
* hypersensitivity to tolvaptan or its excipients
* severe history of allergy (i.e. dyspnea, edema, cutaneous rash…) secondary to any drug administration
* participants with anuria orurinary pathway obstruction (complete or partial)
* natremia ≤133 mmol/l or ≥145 mmol/l
* hypovolemia
* SGOT, SGPT > 1.5 fold upper normal values
* estimated GFR (CKD epi) < 60 ml/min/1.73 m2,)
* current participation to (or being in exclusion period of) another interventional study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-09-06 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
change in serum sodium concentration | Baseline and 6 hours following tolvaptan administration

SECONDARY OUTCOMES:
change in plasma osmolality | Baseline and 6 hours following tolvaptan administration
change urinary sodium excretion | Baseline and 6 hours following tolvaptan administration
change urinary potassium excretion | Baseline and 6 hours following tolvaptan administration
change urinary calcium excretion | Baseline and 6 hours following tolvaptan administration
change urinary magnesium excretion | Baseline and 6 hours following tolvaptan administration
change urinary Acide excretion | Baseline and 6 hours following tolvaptan administration
change urinary chloride excretion | Baseline and 6 hours following tolvaptan administration

CONTACTS AND LOCATIONS:
Overall Officials: Anne BLANCHARD, MD, PhD, Principal Investigator — Assistance Publique des Hopitaux de Paris
Locations (1):
- AP-HP Hôpital Européen Georges Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
IPD underlying published results
Supporting Information: Study Protocol, ICF
Time Frame: One year after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on scientific project and scientific involvement of the PI team.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization.